CLINICAL TRIAL: NCT04574050
Title: A Self - Guided, Internet - Based Intervention for Patients With Chronic Breathlessness (SELF-BREATHE): Feasibility Randomised Controlled Trial
Brief Title: SELF-BREATHE RCT for Chronic Breathlessness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS 285303; 20/LO/1108 (Other: REC / HRA)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Cancer; COPD; Asthma; Bronchiectasis Adult; Interstitial Lung Disease; Cystic Fibrosis; Chronic Heart Failure; Sickle Cell Disease; Renal Failure; Liver Failure; Post COVID-19; Dyspnea
MeSH Terms: conditions — Neoplasms; Pulmonary Disease, Chronic Obstructive; Asthma; Lung Diseases, Interstitial; Cystic Fibrosis; Anemia, Sickle Cell; Renal Insufficiency; Liver Failure; Dyspnea

STUDY DESIGN:
Intervention Model Description: A feasibility RCT comprising two groups:
  1. Intervention (SELF-BREATHE in addition to standard NHS care)
  2. Control group (standard / currently available NHS care)
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SELF-BREATHE (Experimental): Access to a self -guided, internet -based intervention for patients with chronic breathlessness known as SELF-BREATHE
  Interventions: Other: SELF-BREATHE
- Control (No Intervention): standard / currently available NHS care

INTERVENTIONS:
Other: SELF-BREATHE — A self -guided, internet -based intervention for patients with chronic breathlessness
  Arms: SELF-BREATHE

SUMMARY:
A feasibility RCT comprising two groups:

1. Intervention (SELF-BREATHE in addition to standard NHS care)
2. Control group (standard / currently available NHS care)

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age, with the ability to read and type in English
* Access to a computer, or tablet or smart phone, with internet access and the ability to email
* Chronic breathlessness (CB) defined as; breathlessness that persists (>3months) despite optimal pharmacological treatment of the underlying disease including cancer, chronic obstructive pulmonary disease (COPD),asthma, interstitial lung disease (ILD), bronchiectasis, cystic fibrosis (CF) chronic heart failure (CHF), sickle cell disease, chronic renal/ liver failure or post COVID-19
* Chronic breathlessness at rest or on exertion; MRC dysponea score >2
* Willing to engage with short-term self-guided internet-based breathlessness intervention (SELF-BREATHE)
* Able to provide informed consent

Exclusion Criteria:

* Breathlessness of unknown cause
* A primary diagnosis of chronic hyperventilation syndrome
* Currently participating in a rehabilitation programme, e.g. pulmonary/cardiac rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: the number of patients recruited into this study over a 12-month period | 12 months
  The number of patients recruited into this study over a 12-month period

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation TRUST, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No